CLINICAL TRIAL: NCT06510361
Title: A Phase 2 Study of Epcoritamab in Patients With Follicular Lymphoma Not Accomplishing a Complete Response With Upfront Chemoimmunotherapy
Brief Title: Epcoritamab in Patients With Follicular Lymphoma Not Accomplishing a CR With Upfront Chemoimmunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Genmab (Industry)
Responsible Party: Principal Investigator, Gottfried von Keudell, MD PhD, Principle Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-065
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma; Follicular Lymphoma; Lymphoma,Non-Hodgkin; Lymphoma, Non-Hodgkin's, Adult
Keywords: Follicular Lymphoma; Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Non-Hodgkin's, Adult
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Epcoritamab (Experimental): 35 participants will be enrolled and will complete study procedures as follows:
  * Baseline visit with imaging (CT, MRI or PET scan) and bone marrow biopsy.
  * Imaging after Cycles 3 and 6 only.
  * Cycles 1-3:
    --Days 1, 8, 15 and 22 of 28 day cycle: Predetermined dose of Epcoritamab 1x daily
  * Cycles 4-9:
    --Days 1 and 15 of 28 day cycle: Predetermined dose of Epcoritamab 1x daily
  * Cycles 10-12:
    --Day 1 of 28 day cycles: Predetermined dose of Epcoritamab 1x daily
  * End of Treatment visit with imaging and bone marrow biopsy.
  * Follow up: every 3 months for 2 years or until disease worsens.
  * Off study visit with imaging.
  Interventions: Drug: Epcoritamab

INTERVENTIONS:
Drug: Epcoritamab — Humanized IgG1 bispecific antibody, 5 or 60 mL vial, via subcutaneous (under the skin) injection per protocol.
  Other Names: DuoBody-CD3xCD20; GEN3013

SUMMARY:
This research is being done to see if epcoritamab is effective in treating follicular lymphoma as a second line of treatment.

The name of the study drug in this research study is:

-Epcoritamab (a type of antibody)

DETAILED DESCRIPTION:
This is a prospective, phase 2, single arm, open label trial investigating epcoritamab in participants with follicular lymphoma (FL) who have failed to achieve a complete response after frontline therapy. Epcoritamab is a bispecific antibody, a synthetic protein that activates the immune system to target cancer cells.

The U.S. Food and Drug Administration (FDA) has not approved epcoritamab for follicular lymphoma but it has been approved for other uses.

The research study procedures include screening for eligibility, treatment study visits, questionnaires, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, Positron Emission Tomography (PET) scans, electrocardiograms, blood tests, and bone marrow biopsies.

Participants will receive treatment for up to 12 cycles and will be followed for 2 years.

It is expected that about 35 people will take part in this research study.

Genmab, Inc. is funding this research study by providing the study drug, Epcoritamab.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed (fresh or archival tissue) follicular lymphoma grade 1-3A that is CD20+ (by immunophenotype or immunohistochemistry) at time of diagnosis. All degrees of CD20 positivity will be accepted. Composite high-grade lymphoma will be excluded.
* Subjects must have measurable disease at time of enrollment as defined by at least one lymph node with long axis ≥1.5 cm and short axis >1.0 cm and Deauville ≥ 4 seen on baseline PET/CT
* Stage III/IV at initial diagnosis
* 1 prior line (at least 3 cycles) of systemic "upfront" or first-line therapy consisting of anti-CD20 antibody (e.g. obinutuzumab or rituximab) combined with chemotherapy (e.g. bendamustine, CHOP, CVP, or lenalidomide). Rituximab monotherapy, rituximab plus radiation, or radiation alone is not sufficient.
* Subjects need to have achieved a partial response or stable disease as best response following upfront treatment. Subjects with progressive disease will be excluded.
* Subjects must have completed all prior anti-lymphoma therapy at least 4 weeks (28 days) prior to start of epcoritamab.
* Age ≥18 years.
* 3.1.7 Age ≥18 years.
* ECOG performance status ≤ 2
* Life expectancy of greater than 2 years
* Participants must meet the following organ and marrow function as defined below:

  * Absolute neutrophil count ≥1000 cells/mcl (G-CSF allowed if marrow involved with disease)
  * Platelets ≥75,000 cells/mcl (transfusion allowed if marrow involved)
  * Hemoglobin ≥ 8 g/dL (transfusion allowed if marrow involved)
  * Total bilirubin ≤ 1.5 institutional upper limit of normal (ULN). In patients with suspected/known Gilbert's disease total bilirubin up to 3x ULN will be allowed
  * AST(SGOT)/ALT(SGPT) ≤3× institutional ULN unless suspected/known involvement by follicular lymphoma
  * Creatinine ≤ institutional ULN OR creatinine clearance > 45 ml/min (by Cockcroft-Gault estimate or 24-hr creatinine clearance measurement)
* Patients with hepatitis B core antibody positivity with negative PCR on antiviral therapy will be eligible but will be required to receive appropriate antiviral prophylaxis as described in Section 5.4. Patients with Hepatitis C antibody must have undetectable viral load.
* Participants with a history of prior malignancy will be eligible if all treatment of that malignancy was completed at least 2 years prior to enrollment to this study, the treatment was considered "curable-intent", and there is currently no evidence of disease.
* Resolution of toxicities from prior therapy to baseline or grade ≤1 (with the exception of grade 2 peripheral neuropathy or any grade alopecia)
* Ability to understand and the willingness to sign a written informed consent document.
* Females of childbearing potential must agree to practice a highly effective method of birth control (as defined by the EU Clinical Trial Facilitation Group) consistent with local regulations regarding the use of birth control methods for patients participating in clinical trials:

  * Established use of oral, injected or implanted combined (estradiol and progesterone containing) hormonal contraception;
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS);
  * Male partner sterilization (the vasectomized partner should be the sole partner for that patient)
  * True abstinence (when this is in line with the preferred and usual lifestyle of the patient)
* Women must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the trial and for 12 months after receiving the last dose of epcoritamab. Men must also not donate sperm during the trial and for 12 months after receiving the last dose of epcoritamab.
* A man who is sexually active with a woman of childbearing potential must agree to use a barrier method of birth control (i.e. use of condom) during the trial and for 12 months after receiving the last dose of epcoritamab.

Exclusion Criteria:

* Use of investigational agents incorporated into prior induction therapy
* Uncontrolled intercurrent active infection requiring hospitalization or intravenous antimicrobial agents within 4 weeks of start of treatment
* Uncontrolled underlying cardiac conditions including but not limited to congestive heart failure grade III or IV (by NYHA) or EF <45%, unstable angina pectoris, acute myocardial infarction < 6 months, cardiac arrhythmia
* History of uncontrolled neurologic condition including but not limited to seizure disorder, stroke, psychosis, dementia, CNS vasculitis, encephalitis
* EF <45% or need for supplemental O2 at rest to maintain SaO2>89%
* Immunosuppressive therapy for non-lymphoma-related indication within 28 days (or for lymphoma within 10 days) of initiation of treatment, including systemic corticosteroids 10 mg/day or greater of prednisone or equivalent
* Patients with known or suspected CNS involvement or leptomeningeal disease are excluded given concern for potentially increased risk of neurologic toxicity with epcoritamab. Patients with history of CNS malignancy from separate malignancy must have completed CNS-directed therapy and must currently have no evidence of disease
* Pregnant or breastfeeding women or participants unwilling to adhere to institutional guidelines for highly effective contraception for the duration of the therapy are excluded. This is because of the unknown but potential risk of teratogenic or abortifacient effects, as well as potential for adverse events in nursing infants secondary to treatment of the mother, as epcoritamab has not yet been studied in this patient population. A female can be determined to not be of childbearing potential if she meets any of the following criteria:

  * Premenarchal
  * Postmenopausal (>45 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone [FSH] level >40 IU/L or mIU/mL)
  * Permanently sterilized (e.g., bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy)

Note: If the childbearing potential changes after start of the trial (e.g., woman who is not heterosexually active becomes active, premenarchal woman experiences menarche) a woman must begin a highly effective method of birth control, as described under 3.1.15.

* Known current alcohol or drug abuse, psychiatric illness, or unstable social situation that is likely to limit compliance with study requirements
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to epcoritamab
* Exposure to a live or a live attenuated vaccine within 4 weeks
* Patients with HIV will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) | CRR expected to be observed up to 12 months.
  The CRR was defined as the proportion of participants achieving complete response (CR) based on Lugano Response Criteria (Adapted from Cheson, 2014).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | ORR expected to be observed up to 12 months.
  The overall response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on Lugano Response Criteria (Adapted from Cheson, 2014).
Median Progression-Free Survival (PFS) | Survival collected during all visits through 24 months then every 6 months through 5 years.
  Progression-free survival based on the Kaplan-Meier method is defined as the duration between registration and documented disease progression (PD) or death, or is censored at time of last disease assessment.
Median Overall Survival (OS) | Survival observed up to 5 years
  Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Median Time to Next Treatment (TTNT) | Up to 5 years
  TTNT estimated using the Kaplan Meier method is defined as the time from registration until date of initiation of next line of treatment.
Median Duration of Response (DOR) | Observation period up to approximately 12 cycles (1 cycle being 28 days)
  DOR estimated using the Kaplan Meier method, is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) per Lugano Response Criteria, until the first date that recurrent or progressive disease is objectively documented. Participants without progressive disease are censored at the date of last disease assessment.
Median Duration of Complete Response | Observation period up to approximately 12 cycles (1 cycle being 28 days)
  Duration of complete response estimated using the Kaplan Meier method, is measured from the time measurement criteria are met for CR per Lugano Response Criteria, until the first date that recurrent or progressive disease is objectively documented. Participants without progressive disease are censored at the date of last disease assessment.
Rate of Progression of Disease (PD) within 24 months (POD 24) | Up to 24 months
  The POD24 was defined as the proportion of participants achieving progression disease (PD) based on Lugano Response Criteria (Adapted from Cheson, 2014) within 24 months.
Grade 4-5 Treatment-related Toxicity Rate | 12 months (12 cycles of treatment, each cycle is 28 days)
  All grade 4-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 that are not resolved in accordance with treatment guidelines were counted. Rate is the proportion of treated participants experiencing at least one of these adverse events as defined during the time of observation.
Rate of Disappearance of ctDNA | 24 months
  ctDNA assesment done using established method is the proportion of treated participants experiencing disappearance of ctDNA.

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried Von Keudell, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu